CLINICAL TRIAL: NCT03911050
Title: Scavenging of Endogenous Reactive Carbonyl Species by Apple Polyphenols in Healthy Human Subjects
Brief Title: Scavenging of Reactive Carbonyl Species by Apple Polyphenols in Human
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina Agriculture & Technical State University (Other)
Responsible Party: Principal Investigator, Shengmin Sang, Principal Investigator, North Carolina Agriculture & Technical State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 18-0089
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Human Health; Polyphenols; Pharmacokinetics
Keywords: endogenous reactive carbonyl species; apple consumption; formation of carbonyl species adducts of apple polyphenols; pharmacokinetics of adducts in human; intervention
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apple consumption (Experimental): Each subject took apple blends 600 g (made from two apples with seed removal) in a single dose, and samples (urine and blood and feces) at different timepoints were collected following administration of apple blends.
  Interventions: Dietary Supplement: Apple consumption
- Control group (Placebo Comparator): Each subject took breakfast without any apple-related products in a single dose, and samples (urine and blood and feces) at different timepoints were collected following breakfast.
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Apple consumption — Apple blends (600 g) One single dose
  Arms: Apple consumption
Dietary Supplement: Control group — Breakfast without any apple-related products
  Arms: Control group

SUMMARY:
This is an interventional study to investigate formation and pharmacokinetics of reactive carbonyl species adducts of apple polyphenols in human after a single dose of apple consumption.

DETAILED DESCRIPTION:
A crossover design was used. Twelve healthy volunteers were recruited and asked to avoid the consumption of any apple products starting 1 week before intervention and continuing throughout the entire study for a total of 3 weeks.

On week 2, each of six participants received 600 g apple blends (seeds removal) in a single dose, and afterwards, urine and blood samples at different timepoints over 24 h, and fecal sample at different timepoints over 48 h were collected. Meanwhile, other six participants received breakfast (without any apple products) only, and urine and blood samples at different timepoints over 24 h, and fecal sample at different timepoints over 48 h were collected.

On the contrary, on week 3, six participants who received apple blends on week 2 received breakfast only, and six participants who were used as control on week 2 received apple blends. And urine and blood samples at different timepoints over 24 h, and fecal sample at different timepoints over 48 h for both groups were collected.

Samples will be analyzed by LC-MS/MS. Pharmacokinetics of conjugates will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 17 and 30
* Have blood and urine biochemical markers in normal range
* Have no known allergy to apples
* Be not taking antibiotics for six months
* Be not currently taking medication
* Be nonsmoking
* Have no alcoholic intoxication
* Have no extensive exposure to industrial wastes
* Be not frequent charred meat consumption

Exclusion Criteria:

* Individuals with gout
* Individuals with heart diseases
* Individuals with peripheral vascular diseases
* Individuals with degenerative kidney
* Individuals with degenerative liver
* Cancer patients
* Patients with diabetes
* Individuals with GI disorders
* Individuals with endocrine disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Change in urinary levels of reactive carbonyl species (RCS) adducts of apple polyphenols over 24 hours after one single dose of apple consumption | 0-2, 2-4, 4-6, 6-9, 9-12, 12-24 hours post-dose
  Liquid chromatography-tandem mass spectrometry will be utilized to assess RCS adducts of apple polyphenols in urine
Change in plasma levels of RCS adducts of apple polyphenols over 24 hours after one single dose of apple consumption | 0, 0.5, 1, 1.5, 2, 4, 8, 24 hours post-dose
  Liquid chromatography-tandem mass spectrometry will be used to assess RCS adducts of apple polyphenols in plasma
Change in levels of RCS adducts of apple polyphenols in feces over 48 hours after one single dose of apple consumption | 0, 24, 48 hours post-dose
  Liquid chromatography-tandem mass spectrometry will be utilized to assess RCS adducts of apple polyphenols in fecal samples

SECONDARY OUTCOMES:
Change in urinary levels of RCS over 24 hours after one single dose of apple consumption | 0-2, 2-4, 4-6, 6-9, 9-12, 12-24 hours post-dose
  Liquid chromatography-tandem mass spectrometry will be utilized to assess RCS in urine
Change in plasma levels of RCS over 24 hours after one single dose of apple consumption | 0, 0.5, 1, 1.5, 2, 4, 8, 24 hours post-dose
  Liquid chromatography-tandem mass spectrometry will be utilized to assess RCS in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Shengmin Sang, PhD, Principal Investigator — North Carolina Agriculture & Technical State University
Locations (1):
- North Carolina Agriculture and Technical State University, Kannapolis, North Carolina, United States